CLINICAL TRIAL: NCT06706349
Title: Study of Adapted Physical Activity's Impact on Sleep's Quality in Alcohol-use Disorder
Brief Title: Effect of Adapted Physical Activity on Sleep Quality in People With Alcohol Use Disorder
Acronym: APhysOH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/863
Record Dates: First submitted 2024-09-04; First posted 2024-11-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Managed adapted physical activity (Experimental): Participants will receive 3 weekly sessions of supervised adapted physical activity (APA) starting from Visit 3.
  Interventions: Behavioral: APA managed by qualified instructor
- Autonomous adapted physical activity (Placebo Comparator): Participants in this arm will receive a leaflet summarizing WHO recommendations on physical activity at the start of the study.
  Interventions: Behavioral: Autonomous APA

INTERVENTIONS:
Behavioral: APA managed by qualified instructor — Each session will be led by a qualified APA professional and will include a mix of aerobic, anaerobic, and 'mind-body' activities like yoga, tailored to participant preferences. Intensity will range from moderate to vigorous, with activities such as walking, cycling, and club-based exercises for at least 20 minutes per session. Participants will be progressively involved in session planning to support continued practice post-study. Heart rate monitoring will be used during exercises like the 6-minute walk test and chair rise test, while a daily activity calendar will help ensure adherence, documenting session dates, durations, subjective intensity, and activity type.
  Arms: Managed adapted physical activity
Behavioral: Autonomous APA — A leaflet highlighting the importance of non-sedentary behavior according to WHO recommendations will be provided to them. They will have the opportunity to engage in physical activity autonomously according to their preference.
  Arms: Autonomous adapted physical activity

SUMMARY:
This feasibility study aims to assess interest, recruitment, and adherence to a supervised physical activity (APA) program among individuals with Alcohol Use Disorder (AUD). It also investigates the program's impact on sleep quality and efficiency. Key objectives include evaluating recruitment feasibility, assessing randomization acceptance, quantifying adherence rates, and identifying sensitive sleep assessment tools. The study will explore whether APA improves sleep outcomes in AUD patients with sleep complaints, laying groundwork for larger-scale research.

Participants will engage in APA sessions, complete sleep assessments (including sleep diaries and psychometric scales), and provide sociodemographic data and past activity adherence.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 65 years inclusive
* Present an Alcohol Use Disorder (AUD) with at least 2 positive items as defined by the DSM-5
* Present a sleep complaint with a score on the Pittsburgh Sleep Quality Index (PSQI) ≥ 5
* Present active alcohol consumption with at least 6 days of excessive alcohol consumption in the last 4 weeks
* Speak and understand French
* Live within 30 minutes of the University Hospital of Besançon
* Treatment allowed if stabilized for at least 4 weeks
* Signature of informed consent indicating that the subject has understood the purpose and procedures required by the study and agrees to participate and comply with the requirements and restrictions inherent to the study
* Signed automobile safety contract:

  1. The participant agrees to hand over the keys to their vehicle if necessary.
  2. The keys will be returned when the blood alcohol level is below 0.25 mg/L
  3. The participant agrees to name one or more people to contact in case the medical staff deems the participant unfit to return home alone.
* Affiliation to a French social security system or beneficiary of such a system
* Postmenopausal women for at least 24 months, surgically sterilized, or, for women of childbearing age, using an effective method of contraception (oral contraceptives, contraceptive injections, intrauterine devices, double-barrier method, contraceptive patches) (self-reported)

Exclusion Criteria:

* Decompensated heart failure
* Complex ventricular arrhythmias
* Severe uncontrolled hypertension
* Pulmonary hypertension (>60 mmHg)
* Myocarditis or acute pericardial effusion
* Severe obstructive cardiomyopathy
* Severe and/or symptomatic aortic stenosis
* All acute illnesses
* All decompensated or unstable chronic conditions
* Significant malnutrition
* Extreme fatigue and/or manifest physical incapacity
* Severe anemia
* Severe intoxication (psychoactive substances)
* Severe withdrawal syndrome (Cushman >7)
* Relative contraindications for high-intensity physical activities:
* Chronic respiratory insufficiency on long-term oxygen
* Severe chronic respiratory conditions
* Complicated diabetes with severe retinopathy
* Sickle cell disease
* Mild intoxication (psychoactive substances)
* Mild withdrawal syndrome (Cushman >2)
* Musculoskeletal and dermatological limitations: Unhealed traumatic injuries.
* Musculoskeletal and dermatological limitations: Osteoarticular conditions in acute flare (osteoarthritis, arthritis).
* Musculoskeletal and dermatological limitations: Diabetes with plantar ulcer.
* Musculoskeletal and dermatological limitations: Pressure ulcers and evolving or chronic wounds.
* On the day of signing consent: Blood alcohol concentration > 0 mg/L of expired air.
* On the day of signing consent: If blood alcohol concentration is < 0.25 mg/L, the participant may join other therapeutic activities and return home autonomously.
* On the day of signing consent: If blood alcohol concentration is > 0.25 mg/L without clinical signs of intoxication, the participant may join other therapeutic activities and return home accompanied.
* On the day of signing consent: If blood alcohol concentration is > 0.25 mg/L with clinical signs of intoxication, the participant will not join other therapeutic activities. A supervised room placement will be offered, and emergency services may be contacted if intoxication is unusually high (>2 g/L).
* Excessive alcohol consumption ≥ 6 days in the 4 weeks prior to inclusion.
* Average alcohol consumption > 20 g/day or > 100 g/week.
* CIWA score ≥ 9, indicating the need for medication-assisted withdrawal.
* High physical activity levels according to the Global Physical Activity Questionnaire (GPAQ).
* Concurrent treatment with disulfiram, melatonin, and beta-blockers.
* Unstable or recently changed treatments (<4 weeks).
* History of pre-delirium tremens or delirium tremens.
* Substance use disorder (other than alcohol/nicotine per DSM-5).
* Acute psychiatric disorders requiring immediate hospitalization or adjustment of psychotropic medications.
* Advanced somatic disorders contraindicating physical activity.
* Lack of signed automobile safety contract.
* Legal incapacity or refusal to sign consent.
* No health insurance.
* Anticipated poor cooperation or difficulty completing the study
* Pregnant or breastfeeding women.
* Currently in the exclusion period of another study or listed in the national volunteer registry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Sleep duration measured by actigraphy. | Baseline, 6 weeks (midpoint), 12 weeks (end of sessions), and 14 weeks (2 weeks post-intervention)
  Objective measurement of sleep duration (in minutes) using actigraphy over the course of the study.
Circadian parameters measured by urinary melatonin levels. | Baseline, 6 weeks, 12 weeks, and 14 weeks
  Levels of urinary melatonin (in ng/mL) assessed as an indicator of circadian rhythm.
Sleep quality assessed by Pittsburgh Sleep Quality Index (PSQI). | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Subjective sleep quality measured using the PSQI, a validated scale ranging from 0 (better quality) to 21 (poor quality).
Insomnia severity measured by Insomnia Severity Index (ISI). | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Evaluation of insomnia severity using ISI, a composite scale ranging from 0 (no clinically significant insomnia) to 28 (severe insomnia).
Daytime sleepiness assessed by Epworth Sleepiness Scale (ESS). | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Subjective evaluation of daytime sleepiness using ESS, ranging from 0 (no sleepiness) to 24 (severe sleepiness).
Sleep-wake patterns measured by sleep diary. | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Participant-reported data on sleep duration and quality using a daily sleep diary.
Morningness-eveningness preferences measured by Horne and Östberg Scale. | Baseline only.
  Chronotype assessment using the Horne and Östberg Scale, providing a score categorizing participants as morning, intermediate, or evening types.
Adherence to treatment measured by completed APA sessions. | 12 weeks.
  Number of physical activity sessions completed by participants over the course of the study.
Sociodemographic characteristics collected at baseline. | Baseline only.
  Collection of sociodemographic data including age, gender, marital status, education level, and employment status.
Previous adherence to physical activity. | Baseline only.
  Participants' history of engagement in structured physical activity (binary: Yes/No).
Dropout rate during intervention. | 12 weeks.
  Proportion of participants who prematurely discontinued the study intervention.
Impact of personality traits on treatment adherence. | Baseline to 12 weeks.
  Analysis of the relationship between personality traits (assessed by validated scales) and adherence to intervention protocols.

SECONDARY OUTCOMES:
Alcohol Consumption | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Daily alcohol consumption reported in standard units (equivalent to 10g of alcohol) using the Timeline Follow Back (TLFB) method.
Direct Markers of Alcohol Use | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Biological markers directly indicating alcohol consumption.
Indirect Markers of Alcohol Use | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Biological markers indirectly indicating alcohol consumption.
Alcohol Dependence (ADS-Fr Score) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Alcohol dependence evaluated using the French version of the Alcohol Dependence Scale (ADS-Fr).
Alcohol Craving (OCDS Score) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Craving for alcohol assessed using the Obsessive-Compulsive Drinking Scale (OCDS)
Alcohol Craving (VAS Score) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Craving for alcohol assessed using Visual Analog Scales (VAS).
Impact of Craving Profile on Treatment Outcome | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Influence of the craving profile on treatment success analyzed using predefined criteria.
Risk of Transition to Compulsive Exercise (EDS-R Score) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Risk of developing compulsive exercise behaviors evaluated using the Exercise Dependence Scale-Revised (EDS-R).
Physical Capacity (Chair Stand Test) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Functional capacity assessed using the Chair Stand Test.
Physical Capacity (6-Minute Walk Test) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Functional capacity assessed using the 6-Minute Walk Test (6MWT).
Physical Activity Level (GPAQ Score) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Physical activity level measured using the Global Physical Activity Questionnaire (GPAQ).
Physical Activity Level (Physical Activity Calendar) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Physical activity patterns documented using a dedicated physical activity calendar.
Body Mass Index (BMI) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Calculated as weight in kilograms divided by the square of height in meters (kg/m²).
Waist Circumference (WC) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Measurement of waist circumference in centimeters.
Thigh Circumference (TC) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Measurement of thigh circumference in centimeters.
Blood Pressure (BP) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Systolic and diastolic blood pressure measured in millimeters of mercury (mmHg).
Pulse Rate | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Pulse rate measured in beats per minute (bpm).
Depression (QIDS Score) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Depression severity assessed using the Quick Inventory of Depressive Symptomatology (QIDS).
Anxiety (STAI Score) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Anxiety levels evaluated using the State-Trait Anxiety Inventory (STAI).
Impulsivity (UPPS-P Score) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Impulsive behaviors assessed using the UPPS-P Impulsive Behavior Scale.
Self-Esteem (Rosenberg Score) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Self-esteem assessed using the Rosenberg Self-Esteem Scale.
Quality of Life (WHOQOL-BREF Score) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Quality of life assessed using the WHO Quality of Life-BREF (WHOQOL-BREF) questionnaire.
Decision-Making Abilities (MCQ-27 Score) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Decision-making abilities assessed using the Monetary Choice Questionnaire (MCQ-27).
Motivational Abilities (EEfRT Task) | Baseline, 6 weeks, 12 weeks, and 14 weeks.
  Motivational abilities evaluated using the Effort Expenditure for Rewards Task (EEfRT) on a cycle ergometer.

CONTACTS AND LOCATIONS:
Overall Officials: Julie GIUSTINIANI, MD, Principal Investigator — CHU Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No